CLINICAL TRIAL: NCT06135324
Title: Prevalence of Impairments in Cognitive Function and Manual Dexterity in Out-patients With COPD and Associations With Correct Inhaler Techniques (INHALE)
Brief Title: Impairments That Affect Correct Inhaler Use in COPD
Acronym: INHALE
Status: Active, not recruiting | Type: Observational
Sponsor: COPD Foundation (Other)
Collaborators: Viatris Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-INHALE
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: COPD
Keywords: COPD; Inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prevalence of Cognitive impairment and impaired manual dexterity: Determine the prevalence of both cognitive impairment and impaired manual dexterity in stable out-patients with COPD
- Assess relationship of impairments with patient errors using pMDI, SMI, and/or DPIs: assess the relationships of cognitive impairment and impaired manual dexterity with patient errors using their prescribed, current pMDIs, SMIs, and/or DPIs.

SUMMARY:
INHALE is a one-year, multi-site observational research study funded by Viatris, with two aims:

1. Determine the prevalence of both cognitive impairment and impaired manual dexterity in stable out-patients with chronic obstructive pulmonary disease (COPD).
2. Assess the relationship of cognitive impairment and impaired manual dexterity with patient errors using current pMDIs, SMIs and/or DPIs.

DETAILED DESCRIPTION:
To prescribe inhaled therapy for patients with COPD, health care professionals (HCPs) must make three decisions: short vs long-acting medication, medication class (beta2 agonists, muscarinic antagonists and/or corticosteroids) and delivery system.

At present, there is no guidance by national and international groups of experts on selecting the most appropriate delivery system for patients with COPD. On the other hand, there is a general belief among HCPs that there is no difference in efficacy among pressurized metered dose inhalers (pMDIs), slow mist inhalers (SMIs), dry powder inhalers (DPIs), and nebulizer delivery if the patient uses correct inhaler technique. Unfortunately, there is extensive evidence that patients with COPD exhibit numerous errors using hand-held devices. Experts have opined that HCPs should consider prescribing nebulizer medications for patients with COPD based on various factors or conditions, particularly cognitive impairment and problems with manual dexterity. However, there is little if any supportive evidence for these recommendations.

In stable out-patients with an established diagnosis of moderate to very severe COPD (pulmonary function tests within the last 12 months that demonstrate FEV1 < 60% Predicted required for screening purposes), we hypothesize the following:

1. Cognitive impairment (mild to severe) is present in > 20% of this COPD population
2. Impaired manual dexterity (minimally functional to nonfunctional) is present in > 20% of this COPD population
3. Both cognitive impairment and impaired manual dexterity are associated with patient errors using their current hand-held inhalers.

The objectives of this study are:

1. To determine the prevalence of both cognitive impairment and impaired manual dexterity in stable out-patients with COPD
2. To assess the relationships of cognitive impairment and impaired manual dexterity with patient errors using their current pMDIs, SMIs, and/or DPIs.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years
2. > 10 pack-years smoking cigarettes
3. Diagnosis of COPD based on GOLD Criteria
4. Pulmonary function tests showing FEV1 < 60% predicted (pre-BD).
5. Current use of one or more hand-held inhalers (pMDIs, SMIs, and/or DPIs).

Exclusion Criteria:

1. Current diagnosis of dementia or known cognitive impairment -OR-
2. Current diagnosis of impairment in manual dexterity including severe rheumatoid arthritis, severe arthritis/weakness of the hand/wrist, Parkinson's disease, and/or history of a previous cerebral vascular accident (CVA) resulting in significant musculoskeletal deficit (in judgement of PI).

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As this is a novel proposal, there are no data to calculate a sample size. If 20% of patients exhibit cognitive impairment and 20% exhibit impairment in manual dexterity, 500 total patients provide a sample size of at least 100 patients to examine the relationships between these impairments and errors in correct inhaler use. To ensure an adequate number of patients with an impairment, the study team will receive weekly reports containing a summary of proportion of patients exhibiting either cognitive impairment or impairment in manual dexterity and may stop recruitment once at least 100 patients with an impairment and 100 patients with no impairment have been enrolled. A maximum of 500 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence | Through study completion, average of 1 year by assessing cognitive levels using the Mini-Mental State Exam tool and Functional Dexterity Test for impaired manual dexterity function.
  Determine the prevalence of both cognitive impairment and impaired manual dexterity in stable out-patients with COPD.
Errors using inhaler devices | Through study completion, average of 1 year using a standardized check list for assessment of Inhaler Techniques using pMDI, SMI, and/or DPIs.
  Assess the relationships of cognitive impairment and impaired manual dexterity with patient errors using their current pMDIs, SMIs, and/or DPIs.

CONTACTS AND LOCATIONS:
Overall Officials: Donald A Mahler, MD, Principal Investigator — Valley Regional Hospital
Locations (9):
- United States (9):
  - University of Alabama at Birmingham - Lung Health Center, Birmingham, Alabama
  - RUSH University, Chicago, Illinois
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Midwest Chest Consultants, PC, Saint Charles, Missouri
  - Valley Regional Hospital, Claremont, New Hampshire
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Erlanger Health, Chattanooga, Tennessee
  - University of Texas Medical Brach at Galveston, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No